CLINICAL TRIAL: NCT03181659
Title: Therapeutic Exercise and Therapeutic Patient Education With or Without Manual Therapy for Chronic Nonspecific Low Back Pain: a Randomized Control Trial.
Brief Title: Therapeutic Exercise and Therapeutic Patient Education With or Without Manual Therapy for Chronic Nonspecific Low Back Pain.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Roy La Touche Arbizu (Other)
Collaborators: Centro Universitario La Salle (Other); Servicio Madrileño de Salud, Madrid, Spain (Other); Universidad Autonoma de Madrid (Other)
Responsible Party: Sponsor-Investigator, Roy La Touche Arbizu, Centro Superior de Estudios Universitarios La Salle (Universidad Autónoma de Madrid), Universidad Autonoma de Madrid
Organization: Universidad Autonoma de Madrid (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1
Record Dates: First submitted 2017-05-09; First posted 2017-06-09 (Actual); Last update posted 2018-09-06 (Actual); Status verified 2018-09

CONDITIONS: Chronic Nonspecific Low Back Pain; Low Back Pain
Keywords: Musculoskeletal Manipulations; Exercise; Patient Education; Low back pain
MeSH Terms: conditions — Low Back Pain; Motor Activity | interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group 1: patients with NSCLBP who do not seek care (Experimental): Manual Therapy, Therapeutic Education, Therapeutic Exercice
  Interventions: Procedure: Manual Therapy, Therapeutic Education, Therapeutic Exercice
- Group 2: patients with NSCLBP who do not seek care (Experimental): Therapeutic Education, Therapeutic Exercice
  Interventions: Procedure: Therapeutic Education, Therapeutic Exercice
- Group 3: patients with NSCLBP who seek care (Experimental): Manual Therapy, Therapeutic Education, Therapeutic Exercice
  Interventions: Procedure: Manual Therapy, Therapeutic Education, Therapeutic Exercice
- Group 4: patients with NSCLBP who seek care (Experimental): Therapeutic Education, Therapeutic Exercice
  Interventions: Procedure: Therapeutic Education, Therapeutic Exercice

INTERVENTIONS:
Procedure: Manual Therapy, Therapeutic Education, Therapeutic Exercice — They will receive 8 sessions (2 sessions per week) of joint and neural manual therapy, and will receive 4 sessions (1 session per week) of neuroscience education in which mirror therapy and image observation. The therapeutic exercise program is based on stabilization of the lumbopelvic region.
  Arms: Group 1: patients with NSCLBP who do not seek care; Group 3: patients with NSCLBP who seek care
Procedure: Therapeutic Education, Therapeutic Exercice — They will receive a total of 8 sessions (2 sessions per week) of therapeutic exercise based on the stabilization of the lumbopelvic region and will receive 4 sessions (1 session per week) of neuroscience education in which mirror therapy and image observation.
  Arms: Group 2: patients with NSCLBP who do not seek care; Group 4: patients with NSCLBP who seek care

SUMMARY:
This clinical trial study evaluates the effectiveness of a multimodal physiotherapy treatment based on a biobehavioural paradigm in the treatment of non-specific chronic low back pain. The experimental group received treatment based on therapeutic exercise, education in neuroscience, and manual therapy, contrary to the control group, which did not receive manual therapy treatment.

DETAILED DESCRIPTION:
Low back Pain (LBP) is defined by patients as a pain located between the low margins of the costal gridiron and the top limits of the buttock musculature, and it can either be of short or long duration. LBP is the most prevalent musculoskeletal problem, assuming a prevalence between 18,6% and 57,4%. Traditionally, the diagnosis of the DL continues to be based on pathoanatomical criteria even though, in numerous occasions, the outcomes found in complementary tests of image do not correlate with the intensity of pain and the level of disability of the patients. According to the guides of clinical practice, LBP can be divided in three subgroups: firstly, patients whose pain can be associated to a previous pathology, secondly, patients with a diagnosed neuropathic pain associated to a neurological condition, and lastly, patients who present LBP of unspecific characteristics, not preceded by any pathology or relevant damage. According to the World Health Organization, the latter represent 90% of the cases. Thus, this problem supposes a high index of chronicity, and it is the principal reason of labor absenteeism and disability encountered in society, as well as one of the most common motives of consultation in centers of primary care and specialized attention, which results in a high socioeconomic cost. As for the intervention of the CLBP, nowadays there are numerous studies based on disabling the processing of central and peripheral levels of pain by means of a multidisciplinary boarding based on psychology and on a biobehavioral approach. The aim of this study is to evaluate the efficiency of a multimodal treatment by means of therapeutic exercise (TE) and education in neuroscience (NE), with or without manual therapy (MT).

TE is one of the most frequently used techniques, and one of the most effective in patients with CLBP. Research shows reduction of pain in healthy people through either aerobic exercise, resistance exercise, or isometric exercise, showing an increase in pain thresholds and pain intensity. NE aims to change maladaptive beliefs and erroneous thoughts that interfere in the perception of pain and which lead to increase the presence of psychological variables such as fear of movement, hypervigilance, and catastrophism, enhancing the perpetuation and chronicity of the same. Additionally, MT offers a wide range of specific techniques for the treatment of musculoskeletal disorders with the aim of obtaining a modulation of pain through the neurophysiological effects produced at both peripheral and central levels.

The hypothesis of the present study is that TE, when combined with both NE and MT, is more effective on the principal variables of study after 3 months of follow-up. It is a clinical trial randomized with masking of the assessor. An evaluation of the variables previously described will take place, and it will be measured by a trained physical therapist before receiving the treatment. The second evaluation will be conducted after finishing the intervention, whereas a last evaluation will be undertaken after 3 months of follow-up. The intervention will be carried out by a specialized physical therapist that will use a multimodal approach in a simple, randomized way by means of the software known as GraphPad, which allows us to randomly divide the participants into two groups. The group control will receive a treatment based on a total of 8 sessions, at a rate of 2 sessions per week. In total, a number of 4 sessions of NE will take place once per week during a period of four weeks, together with 7 TE sessions. The experimental group will receive the same intervention that the control group in combination with TM based on a protocol, which will develop during a period of 20-25 minutes, 2 sessions per week, in a total of 8 sessions. Groups will have to continue receiving NE and, regularly, they will receive a total of 4 follow-ups on the process of education via audio-visual material.

ELIGIBILITY:
Inclusion Criteria:

* Patients with non specific low back pain lasting for at least 3 months.
* Patients with pain intensity corresponding to at least 3 points on a 10 point analogue visual scale.
* Patients with pain frequency corresponding to at least 10 days per month.
* Men and Women between 18 and 65 years old.

Exclusion Criteria:

* Presence of trauma or surgery to the thoracic or lumbar region.
* Patients with diagnosis of discopathy or radicular symptoms.
* Patients with history of previous physical-therapy intervention for the lumbar region in the last month.
* Any cognitive impairment that hindered viewing of audiovisual material.
* difficulty understanding or communicating.
* Presence of systemic pathology, Central Nervous System or rheumatic disease.
* Inadequate understanding of the Spanish language to follow instructions for measuring and treatment.
* Collaboration of pregnant women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-12-29 (Estimated); Study Completion 2019-05-30 (Estimated)

PRIMARY OUTCOMES:
Disability and function | Change from disability and function at 3 months.
  The Roland Morris Disability Questionnaire (RMDQ) will be used to assess the physical disability in activities of daily living due to low back pain. This self-administered questionnaire consists of 24 items that refer to the limitations of daily activities as a result of low back pain (Roland and Morris, 1983). The total score ranges from 0 to 24 (higher scores indicate a more severe disability level). The Spanish version of RMDQ has been demonstrated as having acceptable psychometric properties (Kovacs et al., 2002).
Pain Intensity | Change from pain intensity at 3 months.
  Pain Intensity will be measured with Visual Analogue Scale (VAS). The VAS consists of a 100-mm line, the left side of which represents "no pain" whereas the right side represents "maximal pain" (Bijur et al., 2001).
Isometric Force Endurance | Change from Isometric force endurance at 3 months.
  To evaluate the force endurance of the lumbar stabilizing muscles, the Ito test is used to test isometric isometric elevation of the trunk (Moreau et al., 2001). This assay was described by Ito et al. 1996 and has a good level of reliability (Ito et al., 1996). In this test the subject will be asked to lie prone on the stretcher. Then, the subject must elevate his head and trunk of the stretcher, in the way that his sternum does not come into contact with it, maintaining the maximum possible cervical flexion. The subjects must maintain this position in the longest possible time, finishing the test after 5 minutes, a state of fatigue or pain appears.

SECONDARY OUTCOMES:
Temporal Summation | Temporal Summation will be assessed up to 1 week before treatment, up to 1 week after treatment and after 3 months of follow up.
  The temporal summation of stimuli will be measured by Von Frey filaments on the area of worst pain in the lumbar region and on the forearm of the non-dominant upper limb as the control area.; At first a single stimulus will be performed on these points, applied for 0.5 seconds, and then the patient will assess the intensity of pain through a VAS scale. Subsequently, on the same points, 10 rhythmic stimuli will be performed at 1-second intervals and again the intensity of pain will be assessed by a VAS (Starkweather et al., 2015).
Two-point discrimination | Two-Point discrimination will be assessed up to 1 week before treatment, up to 1 week after treatment and after 3 months of follow up.
  The discrimination of two points was evaluated both on the healthy side and on the affected side through an ossiometer, which is accountable for measuring the tactile sensitivity. It consists of a small ruler with two mobile tips. During the test the patient was asked to close his eyes while the Physiotherapist produced tactile stimuli through the instrument and the patient indicated whether he felt one or two contacts. Finally, the smallest distance in millimetres recognized by the patient was measured (Catley et al., 2013).
Funcional range | Funcional range will be assessed up to 1 week before treatment, up to 1 week after treatment and after 3 months of follow up.
  The functional range test was developed by Duncan as a predictor of falls in adulthood (Duncan et al., 1990). It is a measure of postural stability from the multi-directional reach of the upper limb with a fixed base. The functional use test was first validated for the former and subsequently for adults obtaining a good reliability of the measurement of stability (Newton et al.,2001) For the calculation of this test, use a measuring device consisting of a tripod containing a rigid tape measure, parallel to the ground, and placed at the height of the acromion of each subject with elbows and hands in complete extension. The subject has to reach as far as possible maintaining the posture for 2-3 seconds without lifting the feet off the ground.
Strength of lumbar region | Strength of the lumbar region will be assessed up to 1 week before treatment, up to 1 week after treatment and after 3 months of follow up.
  The strength of the lumbar region will be measured by a foot dynamometer (Takei TM 5420). The patient should stand on the dynamometer platform with knees extended, elbows extended, hips bent and index fingers holding the bar at knee height. Starting from this position the subject will have to make a previous adjustment of contraction of the musculature of the lumbar region and must perform a movement of lumbar extension. Subjects should maintain contraction for 3 seconds. It is a valid and reliable test to measure the muscular strength of the lumbar region (Coldwells et al.,1994)
Motor control of lumbar region | Motor control will be assessed up to 1 week before treatment, up to 1 week after treatment and after 3 months of follow up.
  Lumbar motor control will be measured by a pressure biofeedback called Stabilizer TM. The measurement protocol in the following procedure; The patient should be supine position with the Stabilizer TM placed in the lumbar region with an initial pressure of 70 mmHg. Then, the patient will be asked to flex the hip and knee at 90 ° with one leg and then with the opposite one repeating the procedure 3 times, then performing a total average. It is a validated and reliable protocol for motor control of the lumbar region (Azevedo et al., 2013)
Range of movement | Range of movement will be assessed up to 1 week before treatment, up to 1 week after treatment and after 3 months of follow up.
  The range of lumbar movement will be measured using a digitized inclinometer based on a mobile application called iHandy ®. Such an application provides the ability to convert the mobile device into an inclinometer. The inclinometer has proven to be a valid and reliable instrument for measuring lumbar range of motion (Saur et al., 1996) The measurement protocol consists of the following process: the patient should stand in a standing position with the arms along the body. The evaluating physiotherapist will mark the T12 level at the height of the last rib and later the L4-L5 level using the iliac crest as the anatomical reference. There will be 5 movements; Thoraco-lumbar flexion, lumbar flexion, thoraco-lumbar extension, right lateral thoraco-lumbar flexion and left lateral thoraco-lumbar flexion (Kolber et al., 2013)
Dynamic Stability | Dynamic Stability will be assessed up to 1 week before treatment, up to 1 week after treatment and after 3 months of follow up.
  Dynamic stability will be assesed with Y-Balance test. It is a reliable clinical test of that evaluates the neuromuscular control of the trunk and the lower limbs (Pilsky et al.2009). The subject is in the center of a three-arm platform, which has one arm in the anterior direction, and two in the posterior direction, one medial and one lateral with a 45º separation between them and 135º with respect to the anterior arm. Each arm has a graphic scale in length measurements for distance measurement. The arm contains a scope aiming objective that the subject will have to slide along the arm to accurately measure how far they can reach with one lower limb while the other is in the center of the platform. Once the maximum possible distance has been reached the subject must pick up his lower limb back to the platform without resting it on the ground. The upper limbs will be supported like a pitcher on the hips
Pain catastrophizing | Pain catastrophizing will be assessed up to 1 week before treatment, up to 1 week after treatment and after 3 months of follow up.
  The Spanish version of the pain catastrophizing scale (PCS) assesses the degree of pain catastrophizing. The PCS has 13 items and a 3-factor structure of rumination, magnification, and helplessness (García Campayo J et al., 2008)
Kinesiophobia | Kinesiophobia will be assessed up to 1 week before treatment, up to 1 week after treatment and after 3 months of follow up.
  Fear of movement or kinesiophobia will be quantified with the Spanish version of the Kinesiophobia Tampa Scale (TSK-11). This instrument demonstrates reliability and validity in patients with chronic pain, being shorter than the original scale. The total score ranges from 11 to 44 points, with the highest scores indicating greater fear of a new injury due to movement (Gómez-Pérez L et al., 2011)
Self-efficacy | Self-efficacy will be assessed up to 1 week before treatment, up to 1 week after treatment and after 3 months of follow up.
  Self-efficacy will be evaluated through the short version of the General Self-Efficacy Scale, which evaluates initiative, persistence, and effort. It is a scale validated in Spanish and has demonstrated validity, reliability and good internal consistency (Herrero et al., 2014)
Anxiety and Depression | Anxiety and Depression will be assessed up to 1 week before treatment, up to 1 week after treatment and after 3 months of follow up.
  Anxiety and Depression will be evaluated through The Spanish version of the Anxiety and Depression Scale (HADS) is a 14-item instrument with a 4-item Likert scale that measures from 0 to 3. This instrument has two subscales consisting of 7 items each (Perez et al.,1995)

CONTACTS AND LOCATIONS:
Locations (1):
- CSEU La Salle, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Roland M, Morris R. A study of the natural history of back pain. Part I: development of a reliable and sensitive measure of disability in low-back pain. Spine (Phila Pa 1976). 1983 Mar;8(2):141-4. doi: 10.1097/00007632-198303000-00004. No abstract available. PMID 6222486
- [Background] Kovacs FM, Llobera J, Gil Del Real MT, Abraira V, Gestoso M, Fernandez C, Primaria Group KA. Validation of the spanish version of the Roland-Morris questionnaire. Spine (Phila Pa 1976). 2002 Mar 1;27(5):538-42. doi: 10.1097/00007632-200203010-00016. PMID 11880841
- [Background] Bijur PE, Silver W, Gallagher EJ. Reliability of the visual analog scale for measurement of acute pain. Acad Emerg Med. 2001 Dec;8(12):1153-7. doi: 10.1111/j.1553-2712.2001.tb01132.x. PMID 11733293
- [Background] Moreau CE, Green BN, Johnson CD, Moreau SR. Isometric back extension endurance tests: a review of the literature. J Manipulative Physiol Ther. 2001 Feb;24(2):110-22. doi: 10.1067/mmt.2001.112563. PMID 11208223
- [Background] Ito T, Shirado O, Suzuki H, Takahashi M, Kaneda K, Strax TE. Lumbar trunk muscle endurance testing: an inexpensive alternative to a machine for evaluation. Arch Phys Med Rehabil. 1996 Jan;77(1):75-9. doi: 10.1016/s0003-9993(96)90224-5. PMID 8554479
- [Background] Starkweather AR, Heineman A, Storey S, Rubia G, Lyon DE, Greenspan J, Dorsey SG. Methods to measure peripheral and central sensitization using quantitative sensory testing: A focus on individuals with low back pain. Appl Nurs Res. 2016 Feb;29:237-41. doi: 10.1016/j.apnr.2015.03.013. Epub 2015 Apr 8. PMID 26856520
- [Background] Catley MJ, Tabor A, Wand BM, Moseley GL. Assessing tactile acuity in rheumatology and musculoskeletal medicine--how reliable are two-point discrimination tests at the neck, hand, back and foot? Rheumatology (Oxford). 2013 Aug;52(8):1454-61. doi: 10.1093/rheumatology/ket140. Epub 2013 Apr 22. PMID 23611918
- [Background] Duncan PW, Weiner DK, Chandler J, Studenski S. Functional reach: a new clinical measure of balance. J Gerontol. 1990 Nov;45(6):M192-7. doi: 10.1093/geronj/45.6.m192. PMID 2229941
- [Background] Newton RA. Validity of the multi-directional reach test: a practical measure for limits of stability in older adults. J Gerontol A Biol Sci Med Sci. 2001 Apr;56(4):M248-52. doi: 10.1093/gerona/56.4.m248. PMID 11283199
- [Background] Coldwells A, Atkinson G, Reilly T. Sources of variation in back and leg dynamometry. Ergonomics. 1994 Jan;37(1):79-86. doi: 10.1080/00140139408963625. PMID 8112285
- [Background] Azevedo DC, Lauria AC, Pereira AR, Andrade GT, Ferreira ML, Ferreira PH, Van Dillen L. Intraexaminer and interexaminer reliability of pressure biofeedback unit for assessing lumbopelvic stability during 6 lower limb movement tests. J Manipulative Physiol Ther. 2013 Jan;36(1):33-43. doi: 10.1016/j.jmpt.2012.12.008. PMID 23380212
- [Background] Saur PM, Ensink FB, Frese K, Seeger D, Hildebrandt J. Lumbar range of motion: reliability and validity of the inclinometer technique in the clinical measurement of trunk flexibility. Spine (Phila Pa 1976). 1996 Jun 1;21(11):1332-8. doi: 10.1097/00007632-199606010-00011. PMID 8725925
- [Background] Kolber MJ, Pizzini M, Robinson A, Yanez D, Hanney WJ. The reliability and concurrent validity of measurements used to quantify lumbar spine mobility: an analysis of an iphone(R) application and gravity based inclinometry. Int J Sports Phys Ther. 2013 Apr;8(2):129-37. PMID 23593551
- [Background] Plisky PJ, Gorman PP, Butler RJ, Kiesel KB, Underwood FB, Elkins B. The reliability of an instrumented device for measuring components of the star excursion balance test. N Am J Sports Phys Ther. 2009 May;4(2):92-9. PMID 21509114
- [Background] Garcia Campayo J, Rodero B, Alda M, Sobradiel N, Montero J, Moreno S. [Validation of the Spanish version of the Pain Catastrophizing Scale in fibromyalgia]. Med Clin (Barc). 2008 Oct 18;131(13):487-92. doi: 10.1157/13127277. Spanish. PMID 19007576
- [Background] Gomez-Perez L, Lopez-Martinez AE, Ruiz-Parraga GT. Psychometric Properties of the Spanish Version of the Tampa Scale for Kinesiophobia (TSK). J Pain. 2011 Apr;12(4):425-35. doi: 10.1016/j.jpain.2010.08.004. PMID 20926355
- [Background] Herrero R, Espinoza M, Molinari G, Etchemendy E, Garcia-Palacios A, Botella C, Banos RM. Psychometric properties of the General Self Efficacy-12 Scale in Spanish: general and clinical population samples. Compr Psychiatry. 2014 Oct;55(7):1738-43. doi: 10.1016/j.comppsych.2014.05.015. Epub 2014 May 28. PMID 24973225